CLINICAL TRIAL: NCT03541759
Title: Pain Management After Elective Shoulder Surgery: A Randomized Quantitative Study Comparing Hydromorphone With Piritramide
Brief Title: Pain Management After Elective Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AUVA Traumazentrum Vienna Site UKH Meidling (Other)
Responsible Party: Principal Investigator, Sandra Boesmueller, MD, PhD, Principal Investigator, AUVA Traumazentrum Vienna Site UKH Meidling
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/18-Anesthesiology
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
Keywords: Elective shoulder surgery, hydromorphone, piritramide
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone; Pirinitramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydromorphone (Active Comparator): Hydromorphone Hcl 4 milligram (mg) Tab 2 times after surgery as basic medication. Hydromorphone Hcl 2.6mg maximum 2 per 24h when numeric rating scale (NRS) > 5.
  Interventions: Drug: Hydromorphone Hcl 4Mg Tab
- Piritramide (Active Comparator): Piritramide 15mg s.c. 2 times after surgery as basic medication. Piritramide 7.5mg s.c. maximum 2 per 24h when numeric rating scale (NRS) > 5.
  Interventions: Drug: Piritramide 15mg s.c.

INTERVENTIONS:
Drug: Hydromorphone Hcl 4Mg Tab — Hydal retard 4Mg Tab 2 times after surgery as basic medication. Hydal retard 2.6Mg maximum 2 per 24h when NRS > 5.
  Other Names: Hydal retard 4Mg
  Arms: Hydromorphone
Drug: Piritramide 15mg s.c. — Dipidolor 15mg s.c. 2 times after surgery as basic medication. Dipidolor 7.5mg s.c. maximum 2 per 24h when NRS > 5.
  Other Names: Dipidolor 15mg s.c.
  Arms: Piritramide

SUMMARY:
Postoperative pain management plays an important role in elective shoulder surgery. The aim of this randomized quantitative study is to compare two frequently used postoperative pain regimes (hydromorphone versus piritramide) regarding onset and duration after the effectiveness of the single-shot interscalene block has diminished.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing elective shoulder surgery with a single-shot interscalene plexus brachialis block in addition to general anesthesia
* patients aged 18-99 years
* patients being capable of giving an informed consent to participation in this study

Exclusion Criteria:

* patients aged below 18 years
* patients with decompensated liver, heart or renal insufficiency
* patients with any kind of lung disease
* patients with a chronic pain syndrome
* patients with a previous pain medication with more than 3 drugs over more than 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Pain management after elective shoulder surgery | 6 months
  Comparison of hydromorphone versus piritramide using the numeric rating scale (NRS; range 0 - 10 points; level 0 representing no pain; level 10 representing the highest pain level)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Steltzer, MD, Prof., Study Chair — Trauma Center Vienna Meidling
Locations (1):
- Austrian Workers Compensation Board Trauma Center Vienna Meidling, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No